CLINICAL TRIAL: NCT02746705
Title: Pilot Study of Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-01189
Record Dates: First submitted 2016-04-04; First posted 2016-04-21 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) (Active Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Cognitive Training Program
- Sham Transcranial Direct Current Stimulation (tDCS) (Sham Comparator)
  Interventions: Device: Sham Transcranial Direct Current Stimulation; Behavioral: Cognitive Training Program

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is a therapeutic development that utilizes low amplitude direct currents to induce changes in cortical excitability. tDCS is expected to produce neuronal polarization of less than one mV (millivolt) 9. tDCS produces relatively diffuse current flow, as demonstrated by imaging studies and computational models
  Other Names: Soterix 1x1 tDCS mini-CT
  Arms: Transcranial Direct Current Stimulation (tDCS)
Device: Sham Transcranial Direct Current Stimulation — During a sham session, the device is programmed to ramp up to the desired intensity (target 2.0 mA) and ramp down for the initial 60 seconds, with no current delivery during the session, and then again at the end of the session. These brief periods of stimulation serve to mimic the effects of a true stimulation session.
  Arms: Sham Transcranial Direct Current Stimulation (tDCS)
Behavioral: Cognitive Training Program

SUMMARY:
This study will test the tolerability and preliminary efficacy of transcranial direct current stimulation (tDCS) combined with a cognitive training program, remotely-delivered using a telemedicine protocol in 60 adults with multiple sclerosis (MS). The study will evaluate the efficacy of tDCS to evaluate two of the most debilitating symptoms of MS: cognitive impairment and fatigue.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) has been demonstrated to:

1. successfully treat fatigue in adults with MS, and
2. improve learning ability and other aspects of cognitive functioning in healthy controls and in participants with a range of medical disorders.

Cognitive impairment in MS remains a major treatment challenge and a trial of tDCS combined with a cognitive training program to treat MS-related cognitive impairment is warranted. However, one barrier for the study of tDCS has been the need for the participant to travel to the study site for each tDCS administration. To address this issue, the biomedical company Soterix, has recently designed a remote-delivery tDCS device designed for use in clinical trials. Therefore, the primary goal of this study is to establish a protocol for remotely-supervised in-home tDCS delivery for studies with MS participants. Established safety and feasibility of remotely-supervised tDCS delivery will facilitate the next steps of larger controlled trials, in both MS as well as other conditions, to determine efficacy and appropriate real-world use.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Definite MS diagnosis, all subtypes [95]
* MS-related changes in cognitive functioning
* A score of 6.5 or lesson the Expanded
* Disability Status Scale (EDSS) OR more than 6.5 with proxy
* Has stable and continuous access to internet service at home compatible with the study laptop (Wi-Fi or ethernet cable)
* Adequate internet capacity for remote monitoring, as tested by http://www.speedtest.net/)
* Adequate home facilities (enough space, access to quiet and distraction free area)
* Able to commit to the two-week period of training sessions with baseline and follow-up visits.
* Able to understand the informed consent process and provide consent to participate in the study

Exclusion Criteria:

* Visual, auditory and motor deficits that would prevent full ability to understand study instructions or operate the tDCS device or study laptop, as judged by treating neurologist or study staff
* Relapse or steroid use in previous month
* History of mental retardation, pervasive developmental disorder or other neurological condition associated with cognitive impairment
* Primary psychiatric disorder that would influence ability to participate
* History of seizures or seizure disorder
* Current chronic headaches or migraines. In addition, if a subject has had a change in the rate or severity of head pressure, headache, or migraine in the past two weeks, they are excluded.
* History of head trauma (e.g., head injury, brain surgery) or medical device implanted in the head (such as Deep Brain Stimulator) or in the neck (such as a Vagus Nerve Stimulator)
* Any skin disorder/sensitive skin (e.g., eczema, severe rashes), blisters, open wounds, burn including sunburns, cuts or irritation, or other skin defects which compromise the integrity of the skin at or near stimulation locations (where electrodes are placed)
* Treatment for a communicable skin disorder currently or over the past 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, Principal Investigator — NYU Langone Medical Center
Locations (1):
- New York University Langone Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Dobbs B, Pawlak N, Biagioni M, Agarwal S, Shaw M, Pilloni G, Bikson M, Datta A, Charvet L. Generalizing remotely supervised transcranial direct current stimulation (tDCS): feasibility and benefit in Parkinson's disease. J Neuroeng Rehabil. 2018 Dec 7;15(1):114. doi: 10.1186/s12984-018-0457-9. PMID 30522497

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Direct Current Stimulation (tDCS): Transcranial Direct Current Stimulation (tDCS): tDCS is a therapeutic development that utilizes low amplitude direct currents to induce changes in cortical excitability. tDCS is expected to produce neuronal polarization of less than one mV (millivolt) 9. tDCS produces relatively diffuse current flow, as demonstrated by imaging studies and computational models
  Cognitive Training Program
- Sham Transcranial Direct Current Stimulation (tDCS): Sham Transcranial Direct Current Stimulation: During a sham session, the device is programmed to ramp up to the desired intensity (target 2.0 mA) and ramp down for the initial 60 seconds, with no current delivery during the session, and then again at the end of the session. These brief periods of stimulation serve to mimic the effects of a true stimulation session.
  Cognitive Training Program
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Transcranial Direct Current Stimulation (tDCS)
Started | 17 | 14
Completed | 15 | 12
Not Completed | 2 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — outlier scores deemed not valid | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Transcranial Direct Current Stimulation (tDCS) | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Customized [Mean (Standard Deviation); unit: years] | 44.8 (16.2) | 43.4 (16.2) | 44.1 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing measures were not administered by the study coordinator due to time limitations at visit. Fatigue assessment was prioritized as primary outcome, while the cognitive measures were collected for exploratory purposes to support power estimates to be used in potential future grant applications.
  Participants
    Female | 8 | 8 | 16
    Male | 7 | 4 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: n=4 total excluded from analyses: n=2 met stop criteria for study procedures, n=1 delayed in completing follow-up, n=1 outlier scores deemed not valid
  Participants
    Black or African American: number analyzed (Participants) | 5 | 4 | 9
    Black or African American | 5 | 4 | 9
    White: number analyzed (Participants) | 10 | 8 | 18
    White | 10 | 8 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Completing at Least 80% of the Targeted Sessions.
Description: 80% is equivalent to n=16 of the targeted 20 transcranial direct current stimulation (tDCS) or sham tDCS sessions.
Time Frame: Four Weeks
Measure: Number; unit: participants
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 15 | 12
participants | 15 | 12

2. Primary Outcome: Change in Total Score of the Brief International Assessment of Cognition in MS (BICAMS)
Description: BICAMS comprises two tests, the Symbol Digit Modalities Test (SDMT) and the Brief Visuospatial Memory Test-Revised (BVMT-R).
  Scoring for SDMT involves summing the number of correct substitutions within the 90 second interval (max = 110. The higher the score, the better).
  Visual/spatial memory is assessed in BICAMS using the BVMTR. In this test, six abstract designs are presented for 10 sec. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. Thus, scores range from 0 to 12 (the higher the score, the better).
  The total score range for BICAMS is 0-122. The higher the score, the better.
Time Frame: Baseline, Four Weeks
Population: 1 participant did not complete this session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 15 | 11
score on a scale | 0.12 (0.47) | 0.29 (0.63)

3. Secondary Outcome: Change in Score on Modified Fatigue Impact Scale (MFIS)
Description: MFIS consists of 21 statements. The number that best indicates how often fatigue has affected the participant in the manner described during the past 4 weeks is circled. Answer choices include: 0 - never, 1 - rarely, 2 - sometimes, 3 - often, 4 - almost always. The total score ranges from 0 to 84. The higher the number, the more frequently fatigue impacted the participant during the past 4 weeks.
Time Frame: Baseline, 4 Weeks
Population: Some participants did not complete the MFIS session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 10 | 9
score on a scale | -11.3 (11.28) | -0.44 (20.81)

4. Secondary Outcome: Change in Score of CogState Brief Battery (CBB)
Description: CBB is a brief, computer-administered cognitive test battery that requires approximately 10 minutes for administration. If the CBB score falls between -10 to +10, it is considered normal. CogState scoring is such that 0 could be considered as performing in the average range for that subtest compared to people of similar age. A negative score means that the performance was lower than average, and a positive score means the performance was higher than average. Higher positive scores (for instance 0.2 becoming 0.5) may indicate slightly better performance and higher negative scores (for instance, -0.4 becoming -0.8) may indicate slightly worsening performance.
Time Frame: Baseline, 4 Week
Population: Some participants did not complete the CBB session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Transcranial Direct Current Stimulation (tDCS)
Number analyzed (Participants) | 14 | 8
score on a scale | -0.02 (0.05) | -0.04 (0.07)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Description: side effect by active and sham participants, with number of participants occurring and total number of occurrences across sessions.
Arm/Group | Transcranial Direct Current Stimulation (tDCS) | Sham Transcranial Direct Current Stimulation (tDCS)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 15/17 | 12/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Direct Current Stimulation (tDCS) (N=17) | Sham Transcranial Direct Current Stimulation (tDCS) (N=14)
Tingling at electrode site (General disorders) | 14 (139) | 11 (104)
Itching at electrode site (General disorders) | 8 (56) | 5 (21)
Heat sensation at electrode site (General disorders) | 8 (63) | 8 (68)
headache (General disorders) | 3 (4) | 3 (11)
Facial muscle twitching (General disorders) | 1 (1) | 0 (0)
Blurred vision (General disorders) | 0 (0) | 1 (1)
Localized head pain (General disorders) | 2 (14) | 1 (2)
Forgetfulness (General disorders) | 2 (2) | 0 (0)
Difficulty concentrating (General disorders) | 2 (2) | 2 (2)
Dizziness (General disorders) | 0 (0) | 1 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT02746705/Prot_SAP_000.pdf